CLINICAL TRIAL: NCT05206279
Title: Laparoscopic Visualization of the Ureters Using Near-infrared Fluorescence After Retrograde Application of Indocyanine Green (ICG) in Deep Infiltrating Endometriosis.
Brief Title: ICG for Visualization of the Ureters in DIE
Acronym: Lavic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Lavic-Trial
Record Dates: First submitted 2021-09-28; First posted 2022-01-25 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Visualization of Ureters in Gynecological Surgery; Deep Infiltrative Endometriosis; ICG (Indocyanine Green); Near Infrared Imaging; Laparoscopy
Keywords: endometriosis; ICG; ureter
MeSH Terms: conditions — Endometriosis | interventions — Cystoscopy

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ureteral ICG injection (Experimental): There is only one arm of the study. All patients will undergo normal laparoscopy. After examining the abdominal structures for presence of endometriosis as well as performing photographic documentation, cystoscopy with intraureteral administration of ICG will be performed, after which intervention the ureters will be examined by laparoscopy. ICG is injected cystoscopy-guided into the ureters (cystoscopy-guided) in a dosage of 5 or 10ml (25mg ICG in 5 or 10ml NaCl) per ureter as a bolus injection.
  Interventions: Drug: Ureteral injection of Indocyanine Green Powder (diluted)

INTERVENTIONS:
Drug: Ureteral injection of Indocyanine Green Powder (diluted) — The intervention we study is the intraureteral injection of ICG during a laparoscopic deep infiltrative endometriosis resection procedure. Cystoscopy with intraureteral administration of ICG will be performed, after which intervention the ureters will be examined by laparoscopy. ICG is injected cystoscopy-guided into the ureters (cystoscopy-guided) in a dosage of 5 or 10ml (25mg ICG in 5 or 10ml NaCl) per ureter as a bolus injection.
  Other Names: Cystoscopy

SUMMARY:
Endometriosis is a common condition with an incidence of approximately 10% of all women in the fertile phase. Deep infiltrating endometriosis (DIE) has been shown to be associated with high morbidity. A retrospective study of 700 patients has shown lower urinary tract involvement in up to 52.6% of cases with DIE. In most studies, the bladder is cited as the most common site of DIE in the urinary tract, with the ureter being the second most common lesion site. In cases of ureteral endometriosis, a procedure called ureterolysis is essential because complete resection of the endometriosis is necessary to resolve or prevent renal obstruction. In addition, ureterolysis is obligatory in the context of dissection of endometriosis involving the rectovaginal septum, sacrouterine ligaments, or rectum. Ureterolysis is the process of freeing the ureter from both endometriotic nodules as a therapeutic procedure and from physiologic surrounding tissue and structures for complete visualization. Because ureterolysis is a high-risk procedure for ureteral lesions, alternatives are desirable.

ICG is a fluorescent dye that has been used for decades for various indications, including retinal angiography, determination of tissue viability, and testing of cardiac and liver function. It has gained an important role in intraoperative visualization of tissue perfusion as well as sentinel lymph nodes in tumor surgery. ICG has also been used and described for ureteral imageability.

However, these studies included small populations of 10-30 patients. None of the aforementioned studies have investigated the imageability of the ureters in endometriosis and with regard to a possible reduction in the need for ureteral dissection.

The investigators perform a cystoscopy with a retrograde injection of ICG in both ureters. ICG and thus the ureters are visualized during laparoscopy by near-infrared light contained in our camera systems. The additional use of fluorescence imaging of the ureters with ICG injected into the ureters during laparoscopic resection of deep infiltrating endometriosis is intended to improve visualization of the ureters and thus may prevent complete ureterolysis, which is considered a high-risk procedure. It is a safe procedure as ICG has been shown to have an excellent safety profile.

The aim of the study is to prove the feasibility of ureteral visualization using intraureteral ICG in 2D laparoscopy for women with deep infiltrating endometriosis by means of near-infrared fluorescence imaging of the ureters.

In our secondary endpoints the investigators want to describe the duration time of ICG injection, the duration until visualization of the ureters, the detection rate of fluorescing ureters after ICG-injection, the duration until maximum fluorescence is achieved, the duration until the ureters can no longer be displayed, the length of performed ureterolysis in centimeters and the safety of intraureteral ICG injection.

DETAILED DESCRIPTION:
Endometriosis is a common illness with an incidence of about 10% of all premenopausal women. Deep infiltrative endometriosis is associated with high morbidity. The resection of deep infiltrative endometriosis may be risky because of the nearby located anatomical structures such as blood vessels, nerves, intestine and ureters, which are exposed for a lesion, especially if involved in the endometriosis. The most common lesions in gynecological surgery are those of the urinary tract. A retrospective study including 213 patients with DIE has shown an affection of the lower urinary tract in DIE in up to 52.6% of cases. Most studies list the bladder as the most common site of urinary tract DIE, with the ureter as the second most common lesion site. In the cases of ureteric endometriosis, an ureterolysis is indispensable as the complete resection of the endometriotic lesions is necessary to resolve or prevent kidney congestion. In addition, the ureterolysis is mandatory in the course of dissection of endometriotic nodules affecting the rectovaginal septum, the sacrouterine ligaments or the rectum. Speaking from ureterolysis the investigators include the procedure of freeing the ureter both from endometriotic nodules as a therapeutic procedure and from physiological surrounding tissue and structures for full visualization. Since the ureterolysis consists in a high-risk procedure for ureteral lesions, alternatives are desirable. Ureteral injuries are among the most feared complications, as they can result in serious consequences such as leakage of urine into the abdomen, congestion of the ureter or kidney and loss of function of the kidney in question. In case of severe ureteral injury, it must be reimplanted in the bladder or an anastomosis must be performed; if this is not possible, a nephrostomy, i.e. direct drainage of urine from the kidney to the outside through the skin, may be necessary. An early diagnosis and possibly already intraoperative therapy by means of suture, insertion of double j catheter or other, is crucial for the prognosis of the ureter and the kidney.

Until now, the preoperative ureteral stent placement has in many hospitals been the standard method for ureteral identification and avoidance of injuries in patients with DIE and imaging-proven involvement of the urinary tract. However, these stents often lead to pain, dysuria and haematuria during the wearing period, which usually lasts several weeks. In gynecologic surgery there is no evidence for the prophylactic ureteral stent placement in order to avoid ureteral injuries.

The investigators investigate if ICG helps to visualize the ureter in laparoscopic operations for deep infiltrating endometriosis and possibly could help prevent complete ureterolysis and thus reducing the risk of lesions to the ureter.

ICG is a fluorescent dye that has been used since 1956 for various indications including retinal angiography, determination of tissue viability, and cardiac and hepatic function testing. It can be used intravenously to visualize vascularization with near-infrared imaging. In the last decade, it has gained an important role in intraoperative visualization of sentinel lymph nodes in tumor surgery and tissue perfusion. ICG has already been used and described for the visualization of the ureters. However, these trials included small populations of 10-30 patients. None of the studies mentioned has investigated the visualization of the ureters in the case of endometriosis and with regard to possibly reducing the necessity of ureteral dissection.

The investigators will perform a retrograde injection of ICG in the ureters during a cystoscopy. ICG and thus the ureters are visualized in laparoscopy through near-infrared light, which is included in our camera systems. The additional use of fluorescence imaging of the ureters with ICG injected into the ureters during a laparoscopic resection of DIE is supposed to improve the visualization of the ureters and therefore may prevent a complete ureterolysis, considered as a high-risk procedure. It's a safe intervention, as ICG has been shown to have an excellent security profile. Allergic reactions, which usually consist of anaphylaxis, have been described extremely rarely. The intraureteral application of ICG has been used clinically and been applied in studies. To date there have been no reports of iatrogenic ureteral injury, perioperative complications or side-effects in patients undergoing the procedure of intraureteral ICG administration. Therefore, the risk of the ureteral administration of ICG is minimal. However, the investigators consider the benefit of a better visualization of the ureters in laparoscopic operations for deep infiltrating endometriosis as substantial.

The aim of the study is to prove the feasibility of ureteral visualization using intraureteral ICG in 2D laparoscopy for women with deep infiltrating endometriosis by means of near-infrared fluorescence imaging of the ureters.

In our secondary endpoints the investigators want to describe the duration time of ICG injection, the duration until visualization of the ureters, the detection rate of fluorescing ureters after ICG-injection, the duration until maximum fluorescence is achieved, the duration until the ureters can no longer be displayed, the length of performed ureterolysis in centimeters and the safety of intraureteral ICG injection.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age 18 or older
* Premenopausal status (menopause is defined as amenorrhea lasting one year or longer)
* Proven (by laparoscopy or MRI) or highly suspected (ultrasound or clinically) deep infiltrating endometriosis

Exclusion Criteria:

* No DIE detectable intraoperatively
* Known or suspected allergy to iodine, shellfish, or ICG dye
* Hyperthyroid metabolic state (excluding treated hyperthyroidism with euthyroid metabolic state)
* Severe renal insufficiency (GFR < 30ml/min)
* Simultaneous therapy with beta-blockers
* Pregnant (positive human chorionic gonadotropin in the blood) or breastfeeding women
* Intention to become pregnant during the course of the study
* Inability to follow the procedures of the study (due to language problems, psychological disorders, dementia)
* Previous history of radiation therapy of the pelvis
* Presence of medical conditions contraindicating general anesthesia or standard laparoscopic surgery
* Active, non treated urinary tract infection
* Active pyelonephritis
* Women having undergone surgery for reimplantation of the ureters (UCNS) or nephrostomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of visualization of the ureters by means of ICG / near-infrared-imaging technique | The injection will take place during surgery, the time frame concerning feasibility corresponds to the duration of the surgery (1 up to 500 minutes)
  The feasibility of the visualization (yes/no) of the ureters using near-infrared fluorescence after retrograde application of ICG into the ureters in patients with suspected or proven deep infiltrating endometriosis undergoing laparoscopy.

SECONDARY OUTCOMES:
Duration time of ICG injection | The time frame corresponds to the whole time of cystoscopy (1 up to 30 minutes)
  The duration time of cystoscopy and ICG injection will be measured
Duration until visualization of ureters | The time frame corresponds to the time from the injection of ICG into the ureters until a laparoscopic visualization of the ICG-stained ureters with near infrared imaging technique (1 up to 500 minutes)
  The duration until visualization of ureters will be measured
Detection rate of fluorescing ureters after ICG-injection | The ureters will be checked for fluorescence immediately after the ICG-injection and then regularly until the end of operation (1 up to 120 minutes)
  During laparoscopic surgery with near infrared imaging after having injected ICG in both ureters, the ureters will be repeatedly checked for fluorescent staining. The detectable (fluorescent) ureters as well as the not detectable (not fluorescent) ureters will be counted and a detection rate of fluorescing ureters after ICG-injection will be calculated
Duration until the ureters can no longer be displayed | The time frame corresponds to the time between visualization of fluorescent ureter until the ureter can no longer be displayed by means of fluorescence in near infrared imaging (1 up to 500 minutes)
  The duration until the ureters can no longer be displayed will be measured during surgery
The length and duration of performed ureterolysis in centimeters | The time frame corresponds to the duration of performed ureterolysis (30 up to 150 Min.)
  The length of performed ureterolysis in centimeters will be measured with the help of a surgical grasping instrument (of the width of 5 millimeters) (1 up to 20cm).

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Siegenthaler, PD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liapis A, Bakas P, Giannopoulos V, Creatsas G. Ureteral injuries during gynecological surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(6):391-3; discussion 394. doi: 10.1007/pl00004045. PMID 11795643
- [Background] Siddighi S, Yune JJ, Hardesty J. Indocyanine green for intraoperative localization of ureter. Am J Obstet Gynecol. 2014 Oct;211(4):436.e1-2. doi: 10.1016/j.ajog.2014.05.017. Epub 2014 May 14. PMID 24835212
- [Background] Ianieri MM, Della Corte L, Campolo F, Cosentino F, Catena U, Bifulco G, Scambia G. Indocyanine green in the surgical management of endometriosis: A systematic review. Acta Obstet Gynecol Scand. 2021 Feb;100(2):189-199. doi: 10.1111/aogs.13971. Epub 2020 Sep 7. PMID 32895911
- [Background] Mandovra P, Kalikar V, Patankar RV. Real-Time Visualization of Ureters Using Indocyanine Green During Laparoscopic Surgeries: Can We Make Surgery Safer? Surg Innov. 2019 Aug;26(4):464-468. doi: 10.1177/1553350619827152. Epub 2019 Feb 8. PMID 30734638
- [Background] Knabben L, Imboden S, Fellmann B, Nirgianakis K, Kuhn A, Mueller MD. Urinary tract endometriosis in patients with deep infiltrating endometriosis: prevalence, symptoms, management, and proposal for a new clinical classification. Fertil Steril. 2015 Jan;103(1):147-52. doi: 10.1016/j.fertnstert.2014.09.028. Epub 2014 Oct 28. PMID 25439849